CLINICAL TRIAL: NCT01156467
Title: Neurally Adjusted Ventilatory Assist (NAVA) in Ventilatory Care of Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Merja Ålander, MD, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EETTMK:26/2010
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Ventilation
Keywords: Neurally adjusted ventilatory assist NAVA; Premature infant; Edi-signal
MeSH Terms: conditions — Respiratory Aspiration; Premature Birth | interventions — Interactive Ventilatory Support; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Infants randomised to this arm will receive a regular nasogastric tube, and the ventilatory care is given as routinely is done.
  Interventions: Device: Control group, ventilation with i-Servo or Stephanie
- NAVA (Active Comparator): Infants randomised to this arm will receive and Edi-catheter as an oro-/nasogastric tube and the Edi-signal will be monitored and when possible NAVA-ventilation used.
  Interventions: Device: Neurally adjusted ventilatory assist, i-Servo, Maquet Nordic (Solna, Sweden)

INTERVENTIONS:
Device: Neurally adjusted ventilatory assist, i-Servo, Maquet Nordic (Solna, Sweden) — Treatment with Edi-catheter
  Arms: NAVA
Device: Control group, ventilation with i-Servo or Stephanie — Ventilatory support is given as routinely is done in the neonatal intensive care unit, with the ventilators available. Normal nasogastric tube is used.
  Arms: Control

SUMMARY:
The purpose of this study is to find out, whether it is possible to improve the ventilatory care of premature infants by using Neurally adjusted ventilatory assist (NAVA).

The study hypothesis is that by using NAVA-technology and/or by monitoring Edi-signal (the electrical signal of diaphragm), it is possible to accomplish ventilatory care to premature infants more individually.

DETAILED DESCRIPTION:
Asynchrony means that the timing of support given by the ventilator is different from patients own breathing pattern. Asynchrony during ventilatory care may increase the risk for complications especially in premature infants with immature lungs.

In this study investigators will compare currently used ventilation methods to a new neurally adjusted ventilatory assist (NAVA). The aim is to find out, whether by using this new method it is possible to decrease the complications associated to ventilatory care and to shorten the need for mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* All children of postconceptional age from 28+0 to 36+6 weeks needing mechanical ventilation for at least 60 minutes

Exclusion Criteria:

* severe birth asphyxia, malformations, chromosomal abnormality or other condition, which will decrease the length of life
* condition which prevents the positioning of an oro-/nasogastric tube

Max Age: 9 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The duration of mechanical ventilation | 1 hour - 6 weeks

SECONDARY OUTCOMES:
Complications associated to mechanical ventilation | 1 hour - 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Timo Saarela, MD, PhD, Study Director — Oulu University Hospital; Merja Ålander, MD, Principal Investigator — Oulu University Hospital
Locations (1):
- University hospital of Oulu, Oulu, North Ostrobothnia, Finland